CLINICAL TRIAL: NCT01683825
Title: Imaging Cardiac Amyloidosis: A Pilot Study Using F-18 Florbetapir Positron Emission Tomography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sharmila Dorbala, Director of Nuclear Cardiology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P001322
Record Dates: First submitted 2012-09-04; First posted 2012-09-12 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Amyloidosis
Keywords: Amyloidosis; Cardiac; Heart; Imaging; Diagnosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- F-18 florbetapir PET-Amyloid Subjects (Experimental): Individuals with documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  Interventions: Drug: F-18 florbetapir PET
- F-18 florbetapir PET-Healthy Controls (Other): Individuals without documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  Interventions: Drug: F-18 florbetapir PET
- F-18 florbetapir PET-Amyloid Reproducibility Subjects (Experimental): Some of the individuals with documented cardiac amyloidosis from arm 1 will undergo a second F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET) within 30 days to measure reproducibility
  Interventions: Drug: F-18 florbetapir PET

INTERVENTIONS:
Drug: F-18 florbetapir PET — Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
  Other Names: F-18 labeled Florbetapir (Trade Name: Amyvid)

SUMMARY:
The primary aim of this pilot study is to determine whether amyloid deposits in the heart can be measured non-invasively by F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET) in 30 individuals with documented cardiac amyloidosis. We will also enroll 15 individuals without cardiac amyloidosis to undergo the F-18 florbetapir imaging as a control group.

The primary hypothesis of this study is that a specific amyloid binding radiotracer will bind to the myocardial amyloid deposits and help quantify cardiac amyloid burden.

A secondary aim of this study is to determine reproducibility of F-18 florbetapir imaging of the myocardium.

DETAILED DESCRIPTION:
F-18 florbetapir has been studied in multiple clinical trials to image beta-amyloid deposition in the brain of subjects with Alzheimers' disease. Florbetapir F-18 has been well tolerated in studies of more than 2000 human subjects. Biodistribution studies in humans revealed predominantly hepatobiliary excretion. The tracer clears rapidly from the blood pool in about 20 minutes. This radiotracer has been recently approved for clinical imaging of brain amyloid in subjects with suspected Alzheimers disease. The investigators propose to test this FDA approved radiotracer for an off label indication in a pilot study to evaluate its potential utility, if any, to image cardiac amyloidosis.

Amyloid related heart disease is associated with LV wall thickening due to infiltration; however, this myocardial wall thickening is not definitively distinguishable from left ventricular myocyte hypertrophy from increased afterload to the heart from hypertension or aortic stenosis. Typically myocardial or other tissue biopsy with typical echo features of amyloidosis is required for confirmation of amyloidosis. This pilot study is designed to understand whether cardiac amyloid burden can be measured using a specific radiotracer targeted against amyloid protein (F-18 Florbetapir). At this point it is unknown of F-18 Florbetapir will bind to either AL or TTR amyloid protein or to both of them or to neither of them. The investigators would like to study 15 patients with AL and 15 patients with TTR amyloidosis to understand these differences if any. The investigators also seek to understand if the signal to noise ratio of the circulating amyloid protein in the blood pool (AL amyloid disease) allows for good differentiation of myocardial amyloid uptake. 15 individuals without cardiac amyloidosis will also be enrolled as controls for this study.

The purpose of the proposed research study is to examine in detail, using quantitative PET, myocardial F-18 Florbetapir uptake in cardiac amyloidosis in order to better understand mechanisms of heart damage in this disease. A secondary aim of this study is to determine reproducibility of F-18 florbetapir imaging of the myocardium in a subset of patients with amyloidosis who return for a second F-18 florbetapir scan within 30 days.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for amyloid subjects:

* Age > 18 years
* Biopsy proven amyloidosis outside the heart with typical echocardiographic appearance of cardiac involvement, or a positive cardiac biopsy.
* Diagnosis of AL amyloidosis by standard criteria (evidence of plasma cell dyscrasia with appropriate tissue staining for AL) OR
* Diagnosis of TTR amyloidosis (no evidence of plasma call dyscrasia and positive TTR staining of amyloid in tissue biopsy)
* Able and willing to provide informed consent to participate in the study procedures

Exclusion Criteria:

* Pregnancy
* Serious non-cardiac medical illness which will preclude research study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03-23 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Dorbala, MBBS, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dorbala S, Vangala D, Semer J, Strader C, Bruyere JR Jr, Di Carli MF, Moore SC, Falk RH. Imaging cardiac amyloidosis: a pilot study using (1)(8)F-florbetapir positron emission tomography. Eur J Nucl Med Mol Imaging. 2014 Sep;41(9):1652-62. doi: 10.1007/s00259-014-2787-6. Epub 2014 May 20. PMID 24841414

RESULTS

PARTICIPANT FLOW:
Groups:
- F-18 Florbetapir PET-Cardiac Amyloidosis Subjects: Individuals with documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
- F-18 Florbetapir PET Cardiac Amyloidosis Reproducibility Arm: Individuals with documented cardiac amyloidosis will undergo two F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET) scans within 30 days.
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
Period: Overall Study
Arm/Group | F-18 Florbetapir PET-Cardiac Amyloidosis Subjects | F-18 Florbetapir PET-Healthy Controls | F-18 Florbetapir PET Cardiac Amyloidosis Reproducibility Arm
Started | 10 | 6 | 7
Completed | 10 | 6 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This table includes baseline data for all 17 amyloidosis subjects including the 7 subjects who underwent a repeat F-18 florbetapir PET/CT scan for reproducibility as baseline characteristics did not change in the short time interval.
Groups:
- F-18 Florbetapir PET- Subjects With Cardiac Amyloidosis: Individuals with documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
- F-18 Florbetapir PET- Controls Without Cardiac Amyloidosis: Individuals without documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
- F-18 Florbetapir PET- Subjects With Cardiac Amyloidosis Reproducibility Arm: Individuals with documented cardiac amyloidosis will undergo two F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET) scans.
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
- Total: Total of all reporting groups
Arm/Group | F-18 Florbetapir PET- Subjects With Cardiac Amyloidosis | F-18 Florbetapir PET- Controls Without Cardiac Amyloidosis | F-18 Florbetapir PET- Subjects With Cardiac Amyloidosis Reproducibility Arm | Total
Number analyzed (Participants) | 10 | 6 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (13.9) | 57.5 (12.2) | 68.1 (5.8) | 64.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 8
  Male | 6 | 5 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 10 | 4 | 5 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 7 | 23
Type of amyloidosis [Count of Participants; unit: Participants]
  Light chain cardiac amyloidosis | 5 | 0 | 7 | 12
  Transthyretin cardiac amyloidosis | 5 | 0 | 0 | 5
  Controls without cardiac amyloidosis | 0 | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Left Ventricular Myocardial F-18 Florbetapir SUVmean
Description: Standardized uptake value (SUV) mean is defined as the mean F-18 florbetapir activity concentration [kBq/ml] measured within the left ventricular myocardial region of interest multiplied by the decay-corrected amount of injected F-18 florbetapir [kBq] normalized to patient weight [g]. In this study we will measure mean left ventricular global myocardial F-18 Florbetapir SUVmean on static images between 4 minutes to 30 minutes post injection of F-18 florbetapir.
Time Frame: 1 day
Population: 10 cardiac amyloidosis subjects, 6 control subjects without cardiac amyloidosis, and 7 subjects with cardiac amyloidosis were included.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- F-18 Florbetapir PET- Controls Without Cardiac Amyloidosis: Control subjects without documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
- F-18 Florbetapir PET-Cardiac Amyloidosis Subjects in Reproducibility Arm: Individuals with documented cardiac amyloidosis will undergo two F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
Arm/Group | F-18 Florbetapir PET-Cardiac Amyloidosis Subjects | F-18 Florbetapir PET- Controls Without Cardiac Amyloidosis | F-18 Florbetapir PET-Cardiac Amyloidosis Subjects in Reproducibility Arm
Number analyzed (Participants) | 10 | 6 | 7
ratio | 3.2 (1.6) | 1.7 (0.9) | 5.0 (1.6)

2. Secondary Outcome: Percent Change in Global Left Ventricular F-18 Florbetapir SUVmean From Scan 1 to Scan 2
Description: We evaluated change in F-18 florbetapir SUVmean from scan 1 to scan 2 as a percentage value [(SUVmean1 minus SUVmean 2)/(SUVmean 1)*100]. In the 7 participants with cardiac amyloidosis who underwent two studies (median of 7 days apart), the percentage change in F-18 florbetapir SUVmean from scan 1 to scan 2 ranged from -38.5% to +20.8% with a median value of +2.24%.
Time Frame: Repeat scan was performed a median of 7 days after baseline study (range 1-46 days)
Population: Subjects with cardiac amyloidosis who underwent two F-18 florbetapir PET/CT scans.
Measure: Mean (Standard Deviation); unit: % change in SUVmean and SD
Groups:
- F-18 Florbetapir PET-Cardiac Amyloidosis Subjects in Reproducibility Arm: Individuals with documented cardiac amyloidosis will undergo F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET).
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
Arm/Group | F-18 Florbetapir PET-Cardiac Amyloidosis Subjects in Reproducibility Arm
Number analyzed (Participants) | 7
% change in SUVmean and SD | 5.65 (19.9)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- F-18 Florbetapir PET-Cardiac Amyloidosis Subjects Reproducibility Arm: Individuals with documented cardiac amyloidosis will undergo two F-18 florbetapir (Trade Name: Amyvid) positron emission tomography (PET) scans within 30 days.
  F-18 florbetapir PET: Cardiac PET images will be obtained following injection of F-18 labeled Florbetapir (Trade Name: Amyvid)
Arm/Group | F-18 Florbetapir PET-Cardiac Amyloidosis Subjects | F-18 Florbetapir PET-Healthy Controls | F-18 Florbetapir PET-Cardiac Amyloidosis Subjects Reproducibility Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/7

LIMITATIONS AND CAVEATS:
The sample size is small. But, cardiac amyloidosis is a rare and under diagnosed disease, it is challenging to enroll more subjects. Also, due to urgency for treatment for AL amyloidosis and changes in heart failure therapy, it was challenging to perform 2 scans without changes in therapy for reproducibility assessment. There is an ongoing competing longitudinal study and most subjects chose to participate in that study, limiting recruitment to this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT01683825/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT01683825/SAP_001.pdf